CLINICAL TRIAL: NCT01865188
Title: An 8-week Randomized, Double-blind, Placebo-controlled Factorial Study to Evaluate the Efficacy and Safety of LCZ696 Alone and in Combination With Amlodipine in Patients With Essential Hypertension
Brief Title: Study of the Efficacy and Safety of LCZ696 Alone and in Combination With Amlodipine in Patients With Hypertension
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLCZ696A2320; 2013-001643-30 (EudraCT Number)
Record Dates: First submitted 2013-05-24; First posted 2013-05-30 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Hypertension
Keywords: LCZ696,; amlodipine,; hypertension,; ABPM
MeSH Terms: conditions — Hypertension | interventions — sacubitril and valsartan sodium hydrate drug combination; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- LCZ696 200 mg (Experimental): Patients randomized to this treatment arm will receive LCZ696 200 mg once daily for 8 weeks.
  Interventions: Drug: LCZ696
- LCZ696 400 mg (Experimental): Patients randomized to this treatment arm will receive LCZ696 400 mg once daily for 8 weeks.
  Interventions: Drug: LCZ696
- Amlodipine 5 mg (Active Comparator): Patients randomized to this treatment arm will receive amlodipine 5 mg once daily for 8 weeks.
  Interventions: Drug: Amlodipine
- Amlodipine 10 mg (Active Comparator): Patients randomized to this treatment arm will receive amlodipine 10 mg once daily for 8 weeks.
  Interventions: Drug: Amlodipine
- LCZ696 200 mg and amlodipine 5 mg (Experimental): Patients randomized to this treatment arm will receive LCZ696 200 mg and amlodipine 5 mg once daily for 8 weeks.
  Interventions: Drug: LCZ696 and amlodipine combination
- LCZ696 200 mg and amlodipine 10 mg (Experimental): Patients randomized to this treatment arm will receive LCZ696 200 mg and amlodipine 5 mg once daily for 1 week followed by LCZ696 200 mg and amlodipine 10 mg once daily for 7 weeks.
  Interventions: Drug: LCZ696 and amlodipine combination
- LCZ696 400 mg and amlodipine 5 mg (Experimental): Patients randomized to this treatment arm will receive LCZ696 200 mg and amlodipine 5 mg once daily for 1 week followed by LCZ696 400 mg and amlodipine 5 mg once daily for 7 weeks.
  Interventions: Drug: LCZ696 and amlodipine combination
- LCZ696 400 mg and amlodipine 10 mg (Experimental): Patients randomized to this treatment arm will receive LCZ696 200 mg and amlodipine 5 mg once daily for 1 week followed by LCZ696 400 mg and amlodipine 10 mg once daily for 7 weeks.
  Interventions: Drug: LCZ696 and amlodipine combination
- Placebo (Placebo Comparator): Patients randomized to this treatment arm will receive placebo once daily for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LCZ696 — Experimental monotherapy doses
  Arms: LCZ696 200 mg; LCZ696 400 mg
Drug: Amlodipine — Active comparator monotherapy doses
  Arms: Amlodipine 10 mg; Amlodipine 5 mg
Drug: LCZ696 and amlodipine combination — Experimental combination doses
  Arms: LCZ696 200 mg and amlodipine 10 mg; LCZ696 200 mg and amlodipine 5 mg; LCZ696 400 mg and amlodipine 10 mg; LCZ696 400 mg and amlodipine 5 mg
Drug: Placebo — Placebo comparator dose
  Arms: Placebo

SUMMARY:
To evaluate the blood pressure lowering effect and safety of LCZ696 when given alone and in combination with amlodipine in patients with essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female outpatients
2. Patients with mild-to-moderate hypertension, untreated or currently taking antihypertensive therapy
3. Treated patients (using antihypertensive treatments within 4 weeks prior to Visit 1) must have an msSBP ≥150 mmHg and <180 mmHg at the randomization visit and msSBP ≥140 mmHg <180 mmHg at the preceding visit.
4. Untreated patients (newly diagnosed with essential hypertension or having a history of hypertension but have not been taking any antihypertensive drugs for at least 4 weeks prior to Visit 1) must have an msSBP ≥150 mmHg and <180 mmHg at both the randomization visit and the preceding visit.
5. Patients must have an absolute difference of ≤15 mmHg in msSBP between the randomization visit and the preceding visit.
6. Ability to communicate and comply with all study requirements and demonstrate good medication compliance (≥ 80% compliance rate) during the treatment run-in period.

Exclusion Criteria:

1. Severe hypertension (msDBP ≥110 mmHg and/or msSBP ≥ 180 mmHg)
2. History of angioedema, drug-related or otherwise
3. History or evidence of a secondary form of hypertension, including but not limited to any of the following: renal parenchymal hypertension, renovascular hypertension (unilateral or bilateral renal artery stenosis), coarctation of the aorta, primary hyperaldosteronism, Cushing's disease, pheochromocytoma, polycystic kidney disease, and drug-induced hypertension
4. Transient ischemic cerebral attack (TIA) during the 12 months prior to Visit 1 or any history of stroke
5. History of myocardial infarction, coronary bypass surgery or any percutaneous coronary intervention (PCI) during the 12 months prior to Visit 1
6. Pregnant or lactating women
7. Women of child-bearing potential not using highly effective methods of contraception Other protocol defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in mean sitting systolic blood pressure (msSBP) of LCZ696 monotherapy compared to placebo | baseline, 8 weeks
  Sitting blood pressure will be measured at trough (immediately prior to dosing at clinic) and recorded at all study visits. At the first study visit, blood pressure will be measured in both arms and the arm with highest sitting SBP will be found and used for all subsequent readings throughout the study. The 4 repeat sitting measurements will be made at 2 minute intervals and the mean of these four sitting systolic blood pressure measurements will be used as the mean sitting systolic blood pressure for that visit.
Change from baseline in mean sitting systolic blood pressure (msSBP) of the combination of LCZ696 and amlodipine compared to LCZ696 and amlodipine alone. | baseline, 8 weeks
  Sitting blood pressure will be measured at trough (immediately prior to dosing at clinic) and recorded at all study visits. The 4 repeat sitting measurements will be made at 2 minute intervals and the mean of these four sitting systolic blood pressure measurements will be used as the mean sitting systolic blood pressure for that visit.

SECONDARY OUTCOMES:
Change from baseline in mean sitting Diastolic Blood Pressure (msDBP) of LCZ696 monotherapy compared to placebo | baseline, 8 weeks
  Sitting blood pressure will be measured at trough (immediately prior to dosing at clinic) and recorded at all study visits. The 4 repeat sitting measurements will be made at 2 minute intervals and the mean of these four sitting diastolic blood pressure measurements will be used as the mean sitting diastolic blood pressure for that visit.
Change from baseline in mean sitting Diastolic Blood Pressure of the combination of LCZ696 and amlodipine compared to LCZ696 and amlodipine alone | baseline, 8 weeks
  Sitting blood pressure will be measured at trough (immediately prior to dosing at clinic) and recorded at all study visits. The 4 repeat sitting measurements will be made at 2 minute intervals and the mean of these four sitting diastolic blood pressure measurements will be used as the mean sitting diastolic blood pressure for that visit.
Change from baseline in pulse pressure | baseline, 8 weeks
  Pulse pressure will be calculated as the difference between msSBP and msDBP for both office BP and ABPM.
Change from baseline in mean 24-hour ambulatory Systolic Blood Pressure of LCZ696 monotherapy compared to placebo | baseline, 8 weeks
  The ABPM cuff will be placed on the non-dominant arm between approximately 7:00 am and 11:00 am and the device will measure blood pressure 3 times per hour for 24 hours.
Change from baseline in mean 24-hour ambulatory Diastolic Blood Pressure of LCZ696 monotherapy compared to placebo | baseline, 8 weeks
  The ABPM cuff will be placed on the non-dominant arm between approximately 7:00 am and 11:00 am and the device will measure blood pressure 3 times per hour for 24 hours.
Change from baseline in mean daytime ( > 6am and ≤ 10 pm) ambulatory Systolic Blood Pressure of LCZ696 monotherapy compared to placebo | baseline, 8 weeks
  The ABPM cuff will be placed on the non-dominant arm between approximately 7:00 am and 11:00 am and the device will measure blood pressure 3 times per hour for 24 hours.
Change from baseline in mean daytime ( > 6am and ≤ 10 pm) ambulatory Diastolic Blood Pressure of LCZ696 monotherapy compared to placebo | baseline, 8 weeks
  The ABPM cuff will be placed on the non-dominant arm between approximately 7:00 am and 11:00 am and the device will measure blood pressure 3 times per hour for 24 hours.
Change from baseline in mean nighttime (> 10 pm and ≤ 6 am) ambulatory Systolic Blood Pressure of LCZ696 monotherapy compared to placebo | baseline, 8 weeks
  The ABPM cuff will be placed on the non-dominant arm between approximately 7:00 am and 11:00 am and the device will measure blood pressure 3 times per hour for 24 hours.
Change from baseline in mean nighttime (> 10 pm and ≤ 6 am) ambulatory Diastolic Blood Pressure of LCZ696 monotherapy compared to placebo | baseline, 8 weeks
  The ABPM cuff will be placed on the non-dominant arm between approximately 7:00 am and 11:00 am and the device will measure blood pressure 3 times per hour for 24 hours.
Change from baseline in trough to peak ratio of mean 24-hour ambulatory Systolic Blood Pressure of LCZ696 monotherapy compared to placebo | baseline, 8 weeks
  The trough to peak ratio of mean 24-hour ambulatory Systolic Blood Pressure will be calculated using the systolic blood pressure effects at trough (post-dosing hour 24) compared to the maximum systolic blood pressure effect found in the hours after dosing.
Change from baseline in trough to peak ratio of mean 24-hour ambulatory Diastolic Blood Pressure of LCZ696 monotherapy compared to placebo | baseline, 8 weeks
  The trough to peak ratio of mean 24-hour ambulatory Diastolic Blood Pressure will be calculated using the diastolic blood pressure effects at trough (post-dosing hour 24) compared to the maximum diastolic blood pressure effect found in the hours after dosing.
Change from baseline in mean 24-hour ambulatory Systolic Blood Pressure of the combination of LCZ696 and amlodipine compared to LCZ696 and amlodipine alone | baseline, 8 weeks
  The ABPM cuff will be placed on the non-dominant arm between approximately 7:00 am and 11:00 am and the device will measure blood pressure 3 times per hour for 24 hours.
Change from baseline in mean 24-hour ambulatory Diastolic Blood Pressure of the combination of LCZ696 and amlodipine compared to LCZ696 and amlodipine alone | baseline, 8 weeks
  The ABPM cuff will be placed on the non-dominant arm between approximately 7:00 am and 11:00 am and the device will measure blood pressure 3 times per hour for 24 hours.
Change from baseline in mean daytime ( > 6am and ≤ 10 pm) ambulatory Systolic Blood Pressure of the combination of LCZ696 and amlodipine compared to LCZ696 and amlodipine alone | baseline, 8 weeks
  The ABPM cuff will be placed on the non-dominant arm between approximately 7:00 am and 11:00 am and the device will measure blood pressure 3 times per hour for 24 hours.
Change from baseline in mean daytime ( > 6am and ≤ 10 pm) ambulatory Diastolic Blood Pressure of the combination of LCZ696 and amlodipine compared to LCZ696 and amlodipine alone | baseline, 8 weeks
  The ABPM cuff will be placed on the non-dominant arm between approximately 7:00 am and 11:00 am and the device will measure blood pressure 3 times per hour for 24 hours.
Change from baseline in mean nighttime (> 10 pm and ≤ 6 am) ambulatory Systolic Blood Pressure of the combination of LCZ696 and amlodipine compared to LCZ696 and amlodipine alone | baseline, 8 weeks
  The ABPM cuff will be placed on the non-dominant arm between approximately 7:00 am and 11:00 am and the device will measure blood pressure 3 times per hour for 24 hours.
Change from baseline in mean nighttime (> 10 pm and ≤ 6 am) ambulatory Diastolic Blood Pressure of the combination of LCZ696 and amlodipine compared to LCZ696 and amlodipine alone | baseline, 8 weeks
  The ABPM cuff will be placed on the non-dominant arm between approximately 7:00 am and 11:00 am and the device will measure blood pressure 3 times per hour for 24 hours.
Percentage of patients achieving msSBP <140 mmHg and msDBP <90 mmHg | 8 weeks
  The percentage of patients achieving blood pressure control (msSBP <140 mmHg and msDBP <90 mmHg) after 8 weeks of treatment will be calculated.
Percentage of patients achieving msSBP <140 mmHg or a reduction ≥20 mmHg from baseline | Baseline, 8 weeks
  The percentage of patients achieving a successful response in msSBP (msSBP <140 mmHg or a reduction ≥20 mmHg from baseline) after 8 weeks of treatment will be calculated.
Percentage of patients achieving msDBP <90 mmHg or a reduction ≥10 mmHg from baseline | Baseline, 8 weeks
  The percentage of patients achieving a successful response in msSBP (msDBP <90 mmHg or a reduction ≥10 mmHg from baseline) after 8 weeks of treatment will be calculated.
Number of patients reporting adverse events | 8 weeks
  As an assessment of safety of monotherapy and combination therapy of LCZ696, total adverse events, serious adverse events and deaths after 8 weeks of treatment will be reported .

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals